CLINICAL TRIAL: NCT02571556
Title: OPEN-LABEL, MULTI-CENTER, PHASE 1b/2a CLINICAL TRIAL DESIGNED TO EVALUATE THE SAFETY AND EFFICACY OF IONTOPHORETIC DEXAMETHASONE PHOSPHATE OPHTHALMIC SOLUTION IN PATIENTS HAVING UNDERGONE CATARACT SURGERY WITH IMPLANTATION OF A POSTERIOR CHAMBER INTRAOCULAR LENS (IOL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGP-437-008
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Patients Having Undergone Unilateral Cataract Extraction and Implantation of a Monofocal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone Phosphate Ophthalmic Solution (Experimental)
  Interventions: Drug: Experimental: Dexamethasone Phosphate Ophthalmic solution (40 mg/mL) delivered by ocular iontophoresis consisting of 4.0 mA-min at 1.5 mA

INTERVENTIONS:
Drug: Experimental: Dexamethasone Phosphate Ophthalmic solution (40 mg/mL) delivered by ocular iontophoresis consisting of 4.0 mA-min at 1.5 mA — Experimental: Dexamethasone Phosphate Ophthalmic solution (40 mg/mL) delivered by ocular iontophoresis consisting of 4.0 mA-min at 1.5 mA
  Other Names: EGP-437

SUMMARY:
To evaluate the safety and efficacy of ocular iontophoresis with dexamethasone phosphate ophthalmic solution, EGP-437®, using the EyeGate® II Drug Delivery System (EGDS) in patients having undergone cataract surgery with implantation of a posterior chamber intraocular lens (IOL)

DETAILED DESCRIPTION:
This will be a Phase 1b/2a, open-label, multi-site study, in which a total of up to 20 eyes of up to 20 patients will be enrolled. Patients having undergone unilateral cataract surgery with implantation of a posterior chamber monofocal intraocular lens (IOL) who are interested in participating in the study will be provided an informed consent form prior to screening. Screening/Baseline procedures which include best corrected visual acuity (BCVA), slit lamp examination, conjunctival injection, and intraocular pressure (IOP) by tonometry will be used to determine eligibility just prior to cataract surgery on Day 0. Eligible subjects will undergo iontophoresis treatment immediately post-cataract surgery on Day 0 and Day 7, and will return to the clinic for examination on Days 1, 14, and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Have undergone unilateral cataract extraction and implantation of a monofocal IOL at the time of enrollment
2. Age 18 to 85 years
3. Receive, understand, and sign a copy of the written informed consent form
4. Be able to return for all study visits and willing to comply with all study-related instructions

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with an anterior chamber cell count of zero on Day 14 | Day 14

SECONDARY OUTCOMES:
The proportion of subjects with a pain score of zero on Day 7 | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided